CLINICAL TRIAL: NCT05451108
Title: A Clinical Trial Evaluating Medical-Grade Polycaprolactone-PCL Pectus Scaffold Implantation With Autologous Fat Grafting for Pectus Excavatum Camouflage
Brief Title: Pectus Excavatum Camouflage
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BellaSeno Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: BellaSeno GmbH (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-PEC-001
Record Dates: First submitted 2022-06-30; First posted 2022-07-11 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Pectus Excavatum
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Insertion of PCL Pectus scaffold (Experimental): Insertion of a custom-made 3D printed medical-grade polycaprolactone (PCL) Pectus scaffold with autologous fat graft for pectus excavatum defect correction.
  Interventions: Device: PCL Pectus Scaffold implantation and autologous fat grafting

INTERVENTIONS:
Device: PCL Pectus Scaffold implantation and autologous fat grafting — A small incision is made in the chest and pre-sternal pocked is defined. Following this, an empty scaffold is implanted at the site of the defect with skin closed directly over it. At the same stage, autologous fat transfer will be performed, harvesting fat from available donor sites such as the thighs and abdomen - depending on scaffold volume and patient morphology. The area will be infiltrated with local anaesthetic tumescent fluid, liposuction performed, and fat transferred to syringes for filtration prior to injection into the scaffold. Fat will not be processed beyond simple filtration to separate liquid from fat to be injected. The scaffold provides structural stability to the chest during the infiltration of the tissue inside the scaffold.

SUMMARY:
The clinical study is testing a new treatment for pectus excavatum called "custom-made 3D printed scaffold-based soft tissue reconstruction". The new method uses a combination of the patients own adipocytes (fat cells) with a 3D printed scaffold (PCL Pectus Scaffold) to support soft tissue regeneration in the patient's chest using the body's natural healing processes.

The implanted scaffold acts as a resorbable frame to support the growth of cells. The substance used for the scaffold is resorbable, it's similar to the substance used for sutures and stitches, and it's already Therapeutic Goods Administration (TGA) approved for bone reconstruction of the skull. The implanted scaffold degrades over time, leaving the tissue in its place.

DETAILED DESCRIPTION:
A 3D printed scaffold made of medical grade polycaprolactone is planned to be implanted to correct pectus excavatum defects. First the patient will be thoroughly evaluated with history taking, examination and medical imaging to determine whether they are suitable for implantation. Imaging will take place as part of the work-up for the trial in the form of a CT scan and MRI. If the patient is deemed suitable for the trial, a custom-made scaffold for the patient chest wall defect is designed based on the medical imaging attained previously. This scaffold is then manufactured and sterilised, before being implanted.

The implantation surgery will be done at a tertiary teaching hospital by an experienced plastic and reconstructive surgeon. During the implantation procedure, the patient's own fat cells are harvested through simple liposuction techniques, usually from the abdomen and thighs depending on the availability of the tissue. The fat cells that are harvested are then injected into the implanted scaffold at the time of implantation. The total length of procedure is estimated to take 1 hour.

The patients progress will be evaluated daily after the procedure while they are in hospital with clinical assessment of the wounds and overall status. On discharge a number of surveys will be performed to document the progress at regular intervals, as well as recurrent MRI studies.

The effectiveness, complications and side-effects will be monitored for up to two years.

All appointments and clinical assessment will be documented in the electronic patient medical record as well as a secure de-identified trial database.

ELIGIBILITY:
Inclusion Criteria:

1. Pectus excavatum defect
2. Patient aged ≥18 and <55 years (patients 55 years and over may still be eligible pending assessment by investigating team and documentation of rationale)
3. Patient willing and able to comply with the study requirements.
4. Patient is eligible to undergo MRI (i.e., no implanted incompatible metal or metal devices, no history of severe claustrophobia).
5. Patient capable of providing valid informed consent.

Exclusion Criteria:

1. Patient with a known history of immunodeficiency including HIV, concomitant systemic corticosteroid therapy, chemotherapy, synchronous haematological malignancy or other cause for secondary/primary immunodeficiency.
2. Patient with known severe concurrent or inter-current illness including cardiovascular, respiratory or immunological illness, psychiatric disorders, alcohol or chemical dependence, possible allergies that would, in the opinion of the Principal Investigator, compromise their safety or compliance or interfere with interpretation of study results.
3. Patient with unstable cardiac or respiratory function due to pectus excavatum or those requiring functional repair.
4. Patients with Body Mass Index (BMI) below 18.5 kg/m2 and above 30 kg/m2. NB: Patients with BMI up to 10% higher than the upper limit (up to 33 kg/m2) can be still enrolled if the treating surgeon confirms that BMI is not associated with any kind of pathology.
5. Patient with polycaprolactone (PCL) allergy
6. Women who are currently pregnant or breast feeding, or who are planning to become pregnant within two years after the pectus excavatum camouflage surgery.
7. Women of childbearing potential without an appropriate contraceptive method.
8. Patient with life expectancy < 36 months.

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of occurrence and type of SADE and AEs related to the surgical procedure or the device (e.g. vital signs, physical exam findings and cardiorespiratory function from baseline to end of study visit) to ensure the safety of device and procedure. | Assessed daily during inpatient stay and at 1-week, at 1-,3-,6-,12-, 24-months and any relevant unscheduled visits post-surgery with 2 years post-surgery being the primary time-point.
  Clinical safety will be assessed by documenting all adverse events regardless of whether they are related to the trial in an adverse events report form - described in detail in the case report form (CRF). These will be carefully evaluated by the principal investigator.

SECONDARY OUTCOMES:
Change in (fat) volume, soft tissue retention and tissue integration from the time of surgery to the end of study visit using radiological and clinical assessments | Assessed pre-surgery and at 1-,3-,6-,12- and 24-months post-surgery.
  Fat volume, soft tissue retention and tissue integration will be evaluated by a senior radiologist utilising serial MRI imaging with assessment of soft tissue volume using a standardised segmentation protocol. Imaging will be taken at regular intervals in conjunction with clinical visits as defined by the protocol.
Change in cardiorespiratory function from baseline to 1 month after surgery | Assessed pre-surgery and at 1-month post-surgery.
  Pre-operative exercise tolerance testing to confirm their suitability for the trial. This will be repeated after complete recovery from the operation (usually after >4 weeks).
  Cardiorespiratory outcome will be assessed using baseline and post-operative cardiopulmonary exercise. Standard Cardio-Pulmonary Exercise Testing (CPET) protocol will be applied and validated by a physician.
Change in pain assessments from baseline to the end of study visit | Assessed pre-surgery, during inpatient stay and at 1-week, at 1-,3-,6-,12- and 24-months and any relevant unscheduled visits post-surgery.
  Pain will be assessed with the numerical pain rating system from 0 (no pain at all) to 10 (worst imaginable pain). It will be tracked in the inpatient setting as well as at post-operative outpatient reviews.
Change in wound healing from the time of surgery to 1 month after surgery | Assessed during inpatient stay and at 1-week and at 1-month post-surgery.
  Wound status will be assessed with the Holger Classification for wounds.
Change in patient quality of life as assessed by Quality of Life (QoL) questionnaires from baseline to the end of study visit | Assessed pre-surgery and at the 3-, 6-, 12- and 24-month clinical reviews.
  The Nuss questionnaire modified for adults (NQ-mA) and the 36-item Short Form Quality of Life (SF-36) questionnaire will be used to assess patient reported functional outcomes from the intervention. A combination of the NQ-mA and the SF-36 questionnaires provides a platform for comparison of the method proposed in this study against the current gold standard surgical management of pectus excavatum, as well as measuring the relative impact on health-related quality of live compared to interventions in other clinical scenarios.

OTHER OUTCOMES:
Observational assessment of health economic measures from the time of surgery to the end of study visit (hospital length of stay, ICU length of stay, operative time, blood loss during surgery (mL)) | Assessed at 24-months post-surgery.
  Length of admission, blood loss during surgery (mL), operative time and complications will be monitored throughout the trial to provide a guide for optimisation of current protocols and potential translation into use of PCL scaffolds for reconstruction in broader clinical settings.
Observational assessment of histological measures following secondary autologous fat graft (AFG) if indicated (general tissue morphology and micropathology, adipose tissue viability, angiogenesis and immune activity) | Assessed at 24-months post-surgery.
  If patients undergo subsequent fat grafting, core biopsy samples will be taken to histologically evaluate the scaffold contents. Specific stains will be used to assess tissue morphology (haematoxylin and eosin and Oli-Red), adipose tissue viability (anti-Perilipin), angiogenesis (anti-von Willebrand Factor/CD 31) and immune activity (M1 and M2 macrophage activity). These data can be correlated with medical imaging, as well as previous data gained from pre-clinical animal models.
Observational and descriptive assessment of clinical photographs, videos and 3D surface scan of the upper torso and chest fields from the time of surgery to the end of study visit | Assessed pre-surgery and at 1-week, at 1-,3-,6-,12- and 24-months post-surgery.
  The aesthetic changes will be evaluated utilising standardised serial pictures, videos and 3D scans with a comparison of the outcome over time. Pictures, videos and 3D scans will be taken at regular intervals in conjunction with clinical visits as defined in the table below.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wagels, Dr, Principal Investigator — Department of Plastic & Reconstructive Surgery Princess Alexandra Hospital
Locations (1):
- Princess Alexandra Hospital - Wooloongabba, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No